CLINICAL TRIAL: NCT06196359
Title: Assessing Function and Pain After Total Knee Arthroplasty With Combined Femoral and Popliteal Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: UHaifa-FPNB
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Total Knee Arthroplasty; Total Knee Replacement; Total Knee Replacement Surgery; Arthritis Knee; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Femoral and Popliteal nerve block (Experimental): Patients who receive a Patients undergoing total knee arthroplasty received a combined femoral and popliteal nerve block (single-shot of each) during the surgical procedure.
  Interventions: Procedure: Combined Femoral and Popliteal nerve block
- Control group (No Intervention): Patients undergoing total knee arthroplasty and didn't receive pain block.

INTERVENTIONS:
Procedure: Combined Femoral and Popliteal nerve block — Patients who receive a combined femoral and popliteal nerve block during surgery, fill out a questionnaire and undergo a muscle strength test before surgery, undergo functional tests, a muscle strength test and are asked about pain intensity after surgery.
  Arms: Combined Femoral and Popliteal nerve block

SUMMARY:
The goal of this interventional study is to examine whether a pain management technique of combined femoral and popliteal nerve block is effective in total knee arthroplasty patients. The main questions it aims to answer are:

Are there differences in postoperative outcomes? Does the nerve block, age, preoperative quadriceps muscle strength and Oxford Knee Score of the patient predict early functional ability? Participants underwent total knee arthroplasty and assessments. Researchers compared pain management techniques to assess effects on postoperative outcomes and identified the importance of preoperative variables a predictors of early functional ability. Further research is required to refine postoperative pain management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Electively assigned for primary knee replacement surgery.
* The American Society of Anesthesiologists physical status score 1-3.

Exclusion Criteria:

* Revision surgery.
* Patients suffering from chronic pain syndrome or chronic opioid use.
* Patients with previous neurological deficits in the lower extremities.
* A cognitive state that does not allow signing of consent or understanding simple instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Timed up & go Test | First day after surgery and third or fourth day after surgery
  Total time to arise from chair, walk 3 m, turn around, return to chair and sit down. Two trials performed and the faster of the two is recorded to the nearest 10th of a second.
Numeric Pain Rating Scale | up to four days after surgery
  An 11-point scale scored from 0 to 10: 0 = no pain, 10= the most intense pain imaginable
Quadriceps Muscle Strength | A 1 day before the surgery, first day after the surgery and third or fourth day after the surgery .
  muscle strength measure by dynamometer (N⋅m)

SECONDARY OUTCOMES:
Elderly Mobility Scale | First day after the surgery and third or fourth day after the surgery
  The Elderly Mobility Scale is a 20 point validated assessment tool for the assessment of frail elderly subjects. The The Elderly Mobility Scale is measured on an ordinal scale of 0-20, when Scores under 10 - generally these patients are dependent in mobility maneuvers; require help with basic activity of daily living, such as transfers, toileting and dressing. Scores between 10 - 13 - generally these patients are borderline in terms of safe mobility and independence in activity of daily living i.e. they require some help with some mobility maneuvers. Scores over 14 - Generally these patients are able to perform mobility maneuvers alone and safely and are independent in basic activity of daily living.
5 Times Sit to Stand Test | First day after the surgery and third or fourth day after the surgery
  The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times.
Hospitalization Duration | At discharge (assessed up to day 10)
  Number of days of hospitalization after the surgery- taken from the pa...
Surgery Duration | During the surgery
  minutes- taken from the patient's file
Consumption of Analgesics | At discharge (assessed up to day 10)
  taken from the patient's file
Occurrence of Falls | At discharge (assessed up to day 10)
  throughout the hospitalization- taken from the patient's file
Oxford Knee Score Questionnaire | A 1 day before the surgery
  The Oxford Knee Score is a patient self-completion patient-reported outcome containing 12 questions on activities of daily living. It provides a single summed score which reflects the severity of problems that the respondent has with their knee. The Oxford Knee Score is scored 0-48 when Score 0-19 May indicate severe knee arthritis. Score 20-29 May indicate moderate to severe knee arthritis. Score 30-39 May indicate mild to moderate knee arthritis. Score 40-48 May indicate satisfactory joint function.

CONTACTS AND LOCATIONS:
Locations (1):
- Galilee Medical Centre, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No